CLINICAL TRIAL: NCT03064529
Title: A Novel Approach to Inpatient Pediatric Physical Activity Measurement - The 6th Vital Sign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Fizan Abdullah, MD, Division Head, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-734
Record Dates: First submitted 2017-02-13; First posted 2017-02-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Surgery; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accelerometer Participants (Experimental): All participants receive an accelerometer to wear around their wrist to measure physical activity continuously beginning 1 week before surgery (when the accelerometer is put on the wrist) and ending 2 weeks after surgery (when the accelerometer is removed from the wrist).
  Interventions: Behavioral: Accelerometer

INTERVENTIONS:
Behavioral: Accelerometer — All participants receive a wrist worn accelerometer to measure physical activity continuously before and after surgery

SUMMARY:
The present study aims to establish the feasibility of the clinical use of 3-axis accelerometers to measure physical activity in hospitalized children after elective surgery.

DETAILED DESCRIPTION:
Purpose:

A nearly universal aspect of hospitalization is a loss of physical activity due to confinement to bed, deconditioning, respiratory compromise, and pain with recovery comprising multifactorial components such as the return to activity, adequate pain control, and overall neurologic function. Assessment of recovery from surgery and the ability to return to full, normal activity has previously been dependent upon subjective clinical evaluation that are subject to observer-to-observer variability, selection bias, or variable interpretation of the qualitative description of movement. Bedside assessments utilizing an accelerometer could change clinical practice by having readily available, quantifiable, reliable and highly accurate data for healthcare providers when they make day-to-day decisions of medical care, as. The present study aims to establish the feasibility of the clinical use of 3-axis accelerometers to measure physical activity in the hospitalized children after abdominal surgery.

Methods:

Participants:

The target study population will be 25 English- or Spanish-speaking children ages 3-18 undergoing elective abdominal surgery with anticipated overnight hospitalization of at least one day. Children must be freely ambulatory without any pre-existing mobility-limitations. Study enrollment and recruitment will occur in Lurie outpatient urology and pediatric surgery clinics over a 6 month period. Parental/guardian consent will be obtained at the preoperative clinical visit.

Accelerometers Actigraph accelerometers (model GT3X; Pensacola, FL) will be obtained from Lurie Consortium to Lower Obesity in Chicago Children (CLOCC). Study participants will be asked to wear accelerometers at the same location throughout the study period unless there is a contraindication to maintain the same location and requires relocation (e.g. interference by IV access). Location preference is the wrist. Patients will wear accelerometers continuously (except for when bathing) for 7 days prior to surgery, the accelerometer will be removed for the operation and placed back on the patient immediately after the operation through 14 days postoperative. Accelerometers will be mailed to children 10 days preoperatively for those whose surgeries are scheduled >2 weeks from preoperative clinic visit along with a return envelop for return of the accelerometer postoperatively; those children who are scheduled for surgery within 2 weeks of their preoperative clinic visit will be provided accelerometers at that clinic visit. Accelerometers will be returned at postoperative clinic visit if within 8 days after surgery or mailed back if postoperative clinic visit is more than 8 days postoperative. Actigraph software will be purchased and will allow preprogramming of accelerometers to begin collection of data 1 week prior to planned surgery date. Reminder phone calls will be placed remind patients to start wearing accelerometers 1 week prior to surgery. Accelerometer movement count data epoch will be measured at 5-second intervals.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-18 undergoing elective surgery with anticipated overnight hospitalization of at least one day

Exclusion Criteria:

* Any children who are non-ambulatory, have any pre-existing mobility limitations, or have a doctor-ordered physical activity limit >48 hours post surgery. Also, patients with surgery scheduled less than 7 days out as protocol calls for the accelerometer to be worn for 7 days pre-surgery

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in physical activity as measured by accelerometer data | Continuous measurement beginning 1 week before surgery (when the accelerometer is placed on the wrist) and ending 2 weeks after (when the accelerometer is removed from the wrist)

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No